CLINICAL TRIAL: NCT05366699
Title: A Randomized Clinical Trial of the LYMPHA Procedure for the Prevention of Lymphedema After Axillary Lymphadenectomy
Brief Title: LYMPHA Procedure for the Prevention of Lymphedema After Axillary Lymphadenectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-53132; NCI-2022-05172 (Other: CTRP); BRS0127 (Other: Stanford OnCore)
Record Dates: First submitted 2022-05-05; First posted 2022-05-09 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Lymphedema, Breast Cancer; Lymphedema
MeSH Terms: conditions — Breast Cancer Lymphedema; Lymphedema

STUDY DESIGN:
Intervention Model Description: After informed consent is obtained, all subjects will undergo an initial study evaluation to establish the pre-operative baseline and to determine eligibility for randomization. Group A will under axillary lymphadenectomy alone, Group B will undergo lymphadenectomy with soft tissue reinforcement(STR), and Group C will undergo axillary lymphadenectomy with immediate lymphatic reconstruction (LYMPHA) using reverse mapping using the SPY System. Each of the baseline measures will be repeated at 3-month intervals over the 12 months of enrollment in the study. These include lymphography, limb volume measurements, skin thickness measurements, bioimpedance spectrosocpy, and quality-of-life assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Other): Group A will under axillary lymphadenectomy alone
  Interventions: Procedure: Axillary lymphadenetomy alone
- Group B (Active Comparator): Group B will undergo axillary lymphadenectomy with soft tissue reinforcement(STR)
  Interventions: Procedure: axillary lymphadenectomy with soft tissue reinforcement
- Group C (Experimental): Group B will undergo axillary lymphadenectomy with immediate lymphatic reconstruction (LYMPHA) using reverse mapping using the SPY System.
  Interventions: Procedure: axillary lymphadenectomy with immediate lymphatic reconstruction (LYMPHA)

INTERVENTIONS:
Procedure: axillary lymphadenectomy with immediate lymphatic reconstruction (LYMPHA) — lymphatic reconstruction where the cut lymphatic vessels are reconstructed by anastamosing to the veins
  Arms: Group C
Procedure: Axillary lymphadenetomy alone — oncologic axillary lymphadenectomy
  Arms: Group A
Procedure: axillary lymphadenectomy with soft tissue reinforcement — axillary lymphadenectomy with soft tissue reinforcement(STR)
  Arms: Group B

SUMMARY:
Lymphedema is a chronic, progressive, and debilitating condition that occurs with disruption or obstruction of the lymphatic system, which commonly occurs a result of breast cancer therapy. The purpose of this study is to determine if the use of a low risk lymphatic reconstruction procedure at the time of axillary lymph node dissection will reduce the risk of developing lymphedema.

Additionally, to determine if this procedure improves objective outcomes of lymphedema and patient quality of life

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 75 years (inclusive)
* Patients undergoing unilateral or bilateral breast cancer related axillary lymphadenectomy
* Free of distant metastasis in preoperative screening
* Histology results of axillary lymph nodes could be either Negative or Positive
* Patients who undergo preoperative chemotherapy can be included
* Willingness and ability to provide written informed consent
* Willingness and ability to comply with all study procedures

Exclusion Criteria:

* Primary lymphedema of the affected upper limb
* Secondary lymphedema of the affected limb prior to the lymphadenectomy
* Radiotherapy at the axilla before the study / surgery
* Allergic reaction to porcine collagen or ICG
* Receiving radiation therapy to the involved nodal basin in a period less than 4 weeks after the surgery
* Concurrent participation in a clinical trial of any other investigational drug or therapy, regardless of indication, within 1 month before screening
* Other medical condition that could lead to limb edema, such as (but not limited to primary lymphedema or acute venous thrombosis
* Other medical condition that could result in symptoms overlapping those of lymphedema in the affected limb (e.g., pain, swelling, decreased range of motion)
* Either of the following, at the time of baseline evaluation: ipsilateral:contralateral limb volume ratio>1.1 or R0 bioimpedance ratio > 1.106 when the nondominant limb is at risk, and 1.134 when the dominant limb is at risk.
* Life expectancy < 2 years for any reason
* Pregnancy or nursing
* Substance abuse (such as alcohol or drug abuse) within 6 months prior to screening
* Severe psychiatric disease
* Significant or chronic renal insufficiency (defined as serum creatinine > 2.5 mg/dL or an estimated glomerular filtration rate [eGFR] < 30 mL/min at screening) or requires dialytic support
* Hepatic dysfunction, defined as alanine transaminase (ALT) or aspartate transaminase (AST) levels > 3 × upper limit of the normal range (ULN) and/or bilirubin level > 2 × ULN at screening
* Absolute neutrophil count < 1500 mm3 at screening
* Hemoglobin concentration < 9 g/dL at screening
* Any reason (in addition to those listed above) that, in the opinion of the investigator, precludes full participation in the study

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-09-10 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Lymphatic flow pattern of whole limb | 2 yr
  In the early lymphedema stages this exam allows to detect percutaneously the lymphatic vessels of the whole limb, up to about 1 cm in depth from the skin surface, by an infrared camera visualization system after intra-dermal injection of ICG in the hand. The change in the lymphatic pattern and reduction in the ICG velocity will be tested to find a correlation with other used diagnostic parameters like volume change and bioimpedance spectroscopy.
Limb Volume | 2 yr
  Limb volume as measured by serial assessment
Skin thickness measurements | 2 yr
  Skin thickness is changed by lymphedema
Bioiimpedance spectroscopy | 2 yr
  Impedance of the skin changes with lymphedema
Quality of life | 2 yr
  Questionnaire to determine patient reported quality of life. Measured by limb-lymphedema-specific quality of life (LYMQOL) tool. The LYMQOL is divided into four domains: Function, Appearance, Symptoms, and Mood, as well as yielding an overall quality-of-life score

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Cancer Institute, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2024-06-13): https://cdn.clinicaltrials.gov/large-docs/99/NCT05366699/Prot_001.pdf
  • Informed Consent Form (2021-06-15): https://cdn.clinicaltrials.gov/large-docs/99/NCT05366699/ICF_000.pdf